CLINICAL TRIAL: NCT06412354
Title: VIVHEART Transcatheter Aortic Valve Replacement (TAVR) Self-centering Catheter First-in-human Feasibility Trial (VIV-FIH)
Brief Title: EasyCrossTM Device-Self-centering Catheter
Acronym: VIV-FIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivheart s.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP01
Record Dates: First submitted 2024-04-30; First posted 2024-05-14 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-05

CONDITIONS: Transcatheter Aortic Valve Replacement (TAVR)

STUDY DESIGN:
Intervention Model Description: The VIVHEART EasyCross™ fist-in human (VIV-FIH) study is a singlecenter, prospective, open-label, non-randomized, single-group assignment, first-in-human feasibility trial of the VIVHEART EasyCross™ catheter used according to the indication of use. The experimental part of the trial which differs from the traditional TAVR procedure is the use of the self-centering catheter from its insertion in an artery and up to its removal from the patient body (henceforth "investigational procedure").
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VIV-FIH (Experimental): The VIVHEART EasyCross™ fist-in human (VIV-FIH) study is a single center, prospective, open-label, non-randomized, single-group assignment, first-in-human feasibility trial of the VIVHEART EasyCross™ catheter used according to the indication of use. The experimental part of the trial which differs from the traditional TAVR procedure is the use of the self-centering catheter from its insertion in an artery and up to its removal from the patient body (henceforth "investigational procedure").
  Interventions: Device: EasyCross™ first-in human

INTERVENTIONS:
Device: EasyCross™ first-in human — At T0 the patient will undergo the TAVR procedure including the investigational procedure with the VIVHEART EasyCross™ catheter.
  The interventional cardiologist will introduce the VIVHEART EasyCross™ catheter through the femoral artery with a percutaneous access according to the clinical practice through a vascular introducer on an already positioned guidewire. An operator in the procedure room will start a chronometer at this point to measure the investigational device crossing procedure duration.
  The VIVHEART EasyCross™ catheter will be progressed into the aorta and up to the aortic valve.
  At that time the external part of the VIVHEART EasyCross™ catheter will be opened to allow the self-centering of the catheter on the aortic valve. The guidewire will be introduced and once having crossed the valve the VIVHEART EasyCross™ catheter will be retracted by the physician and removed from the patient's body.

SUMMARY:
VIVHEART EasyCross™ is a self-centering device for inserting a guidewire through a heart valve. It consists in a temporary catheter inserted into an artery with a terminal part able to expand a distal structure with 6 arms ("basket") to allow distancing of the catheter from the vessels walls and thus facilitating the passage of the guide wire through the aortic valve. The device is expected to reduce the attempts and the time needed to cross the valve and improves the safety of TAVR procedure

DETAILED DESCRIPTION:
VIVHEART EasyCross™ is a self-centering device for inserting a guidewire through a heart valve. It consists in a temporary catheter inserted into an artery with a terminal part able to expand a distal structure with 6 arms ("basket") to allow distancing of the catheter from the vessels walls and thus facilitating the passage of the guide wire through the aortic valve. The device is expected to reduce the attempts and the time needed to cross the valve and improves the safety of TAVR procedure.

EasyCross™ device is a catheter is intended to allow a rapid and safe centering of a heart valve in order to direct and introduce a guidewire through it. The intended purpose is the use of the device during percutaneous TAVR procedures, including TAVR of a native valve, recrossing and balloon post-dilation of a prosthetic aortic valve, or a valve-in-valve aortic valve replacement within the scope of the CE mark.

The VIVHEART EasyCross™ device is intended for patients candidate to TAVR of a native valve, recrossing and balloon post-dilation of a prosthetic aortic valve, or a valve-in-valve aortic valve replacement. The suitability of the patient is to be verified case by case by the specialized physician, by means of proper physical examination and instrumental evaluation, according to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years old
* Candidate to TAVR of a native valve, recrossing and balloon postdilation of a prosthetic aortic valve, or a valve-in-valve aortic valve replacement.
* Willingness to undergo follow-up visits.
* Ability to understand scope, content and risks of the study, and provide informed consent to participation.

Exclusion Criteria:

* Contraindications for endovascular procedures
* Pregnancy or breastfeeding females at screening and at time of investigational procedure
* Hemodynamically unstable or other clinical conditions increasing the risk of transcatheter valve procedure failure
* Needing emergent procedure
* Allergies to components of the device
* Allergies to drugs or contrast material that may be used during the investigational procedure and all the TAVR procedure
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants with AE /SAE linked or no linked with the EasyCross device | Day of procedure; 1 week; 4 week
  The primary endpoint is the safety of VIVHEART EasyCross™ catheter, in term of adverse events (AE) and serious adverse events (SAE). Occurrence of any AE will be recorded, in particular the following AE will be coded and investigated as adverse events of special interest (AESI):
  * Intra-operative death,
  * Any intra-operative complication due to device malfunction,
  * Any embolization event,
  * Any allergic reaction.

SECONDARY OUTCOMES:
Time (in minutes) spent to crossing the valve witn EasyCross device | during procedure
  The secondary endpoints will evaluate the performances of the VIVHEART
  EasyCross™ catheter in terms of:
  - Investigational device crossing procedure duration, assesmed in minutes starting by introduction of Easycross catheter to crossing the valve.

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Scientific Institute, Milan, Italy